CLINICAL TRIAL: NCT05293548
Title: A Randomized, Controlled Clinical Trial on Sequential Immunization of Recombinant COVID-19 Vaccine (CHO Cell, NVSI-06-09) and Inactivated COVID-19 Vaccine (Vero Cell) in Population Aged 18 Years and Above
Brief Title: A Clinical Trial on Sequential Immunization of Recombinant COVID-19 Vaccine (CHO Cell, NVSI-06-09) and Inactivated COVID-19 Vaccine (Vero Cell)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: China National Biotec Group Company Limited (Industry); Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CNBG-REC-2022002
Record Dates: First submitted 2022-03-22; First posted 2022-03-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVSI-06-09 Sequential Immunization Group (Experimental): the subjects who have been vaccinated with 2 doses/3 doses of inactivated COVID-19 vaccine (Vero cell) for ≥6 months
  Interventions: Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-09)
- Inactivated Vaccine Sequential Immunization Group (Active Comparator): the subjects who have been vaccinated with 2 doses/3 doses of inactivated COVID-19 vaccine (Vero cell) for ≥6 months
  Interventions: Biological: Inactivated COVID-19 vaccine (Vero cells)

INTERVENTIONS:
Biological: Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-09) — Intramuscular injection of Recombinant COVID-19 Vaccine (CHO cell，NVSI-06-09) in the deltoid muscle of the upper arm
  Arms: NVSI-06-09 Sequential Immunization Group
Biological: Inactivated COVID-19 vaccine (Vero cells) — Biological/Vaccine: Inactivated COVID-19 vaccine (Vero cells) Intramuscular injection of Inactivated COVID-19 vaccine (Vero cells) in the deltoid muscle of the upper arm
  Arms: Inactivated Vaccine Sequential Immunization Group

SUMMARY:
A total of 516 healthy subjects aged 18 years and above who have been vaccinated with 2 doses/3 doses of inactivated COVID-19 vaccine, will be enrolled, and randomly assigned to experimental group and control group in a 1:1 ratio, with 258 subjects in each sequential group.

ELIGIBILITY:
Inclusion Criteria:

* Age: population aged 18 years and above;
* Judged by the investigator that the health condition is well after inquiry and physical examination;
* Vaccinated with 2 or 3 doses of inactivated COVID-19 vaccine (Vero Cell vaccine) 6 months prior to study screening and according to product insert;
* Female participants who are not pregnant or nursing or at the time of enrolment (confirmed via negative urine pregnancy test), and do not have plans to become pregnant within the first 6 months after enrollment. Effective contraceptive measures have been taken within 2 weeks before study inclusion and initiation;
* Be able and willing to provide written informed consent to participate in the study and complete all study requirements according to the study protocol;

Exclusion Criteria:

* COVID-19 infection positive patients (including suspected or asymptomatic cases);
* Have a history of SARS and MERS infection;
* Have been vaccinated by any COVID-19 Vaccines other than Vero Cell vaccine；
* Have an axillary temperature 37.3 (forehead temperature 37.8℃℃);
* Have had previous allergic reactions to vaccination (such as acute allergic reactions, urticaria, eczema, dyspnea, angioneurotic oedema or abdominal pain) or allergy to known components of COVID-19 vaccine;
* History of thrombocytopenia or other coagulation disorders;
* Patients with known immunological impairment or immunocompromised.
* Received whole blood, blood products, plasma and/or immunoglobulin therapy within 3 months before study enrollment
* Have known or suspected severe illness such as respiratory illness, acute infection or active attacks of chronic illness, liver and kidney disease, severe diabetes mellitus, malignant tumour, infectious or allergic skin disease, human immunodeficiency virus (HIV) infection (test report available);
* Diagnosed with serious cardiovascular diseases such as cardiopulmonary failure, drug-uncontrolled hypertension (Systolic blood pressure 160 mmHg and/or diastolic blood pressure 95 mmHg).
* Received live attenuated vaccines within 1 month before study enrollment;
* Received inactivated vaccines within 14 days before study enrollment;
* Received other investigational drugs within 6 months before study enrollment;
* Other vaccination-related contraindications considered by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
GMT (Omicron) of anti-SARS-CoV-2 neutralizing antibody in adults ≥18 years of age | 14 days after sequential immunization of one booster dose
the 4-fold rise rate of anti-omicron neutralizing antibody in adults ≥18 years of age | 14 days after a single dose of the booster vaccine
The incidence rate of any adverse reactions/events | within 30 minutes after vaccination
The incidence severity of any adverse reactions/events | within 30 minutes after vaccination
The incidence rate of solicited adverse reactions/events | within 0-7 days after vaccination
The incidence severity of solicited adverse reactions/events | within 0-7 days after vaccination
The incidence rate of solicited adverse reactions/events | within 8-30 days after vaccination
The incidence severity of solicited adverse reactions/events | within 8-30 days after immunization
The incidence of SAE observed | up to 12 months after full course of immunization
The incidence of AESI observed | up to 12 months after full course of immunization

SECONDARY OUTCOMES:
4-fold rise rate of anti-omicron neutralizing antibody in adults ≥18 years of age | 28 days after sequential immunization of one booster dose
GMT of anti-omicron neutralizing antibody in adults ≥18 years of age | 28 days after sequential immunization of one booster dose
4-fold rise rate of anti-SARS-CoV-2 neutralizing antibody in adults ≥18 years of age | 28 days after sequential immunization of one booster dose
GMT of anti-omicron IgG antibody in adults ≥18 years of age | before booster vaccination and 28 days after a single dose of the booster vaccine
4-fold rise rate of anti-omicron IgG antibody in adults ≥18 years of age | before booster vaccination and 28 days after a single dose of the booster vaccine
proportions of neutralizing antibody tittered 1: 16, 1: 32 and 1: 64 of anti-SARS-CoV-2 IgG antibody in adults ≥18 years of age | before booster vaccination and 28 days after a single dose of the booster vaccine
GMI of anti-omicron IgG antibody in adults ≥18 years of age | before booster vaccination and 28 days after a single dose of the booster vaccine
GMTs of anti-omicron neutralizing antibody | 3 months, 6 months, 9 months and 12 months after sequential immunization
IgG antibody of anti-omicron neutralizing antibody | 3 months, 6 months, 9 months and 12 months after sequential immunization
the proportions of neutralizing antibody titered 1: 16, 1: 32 and 1: 64 | 3 months, 6 months, 9 months and 12 months after sequential immunization

OTHER OUTCOMES:
The efficacy of recombinant COVID-19 vaccine (CHO cell, NVSI-06-09) against COVID-19, severe cases and deaths after 14 days following sequential immunization in adults ≥18 years of age | During the study，an average of one and a half years
Cross-protecting effect of neutralizing antibodies against different variants (Alpha, Beta, Delta, and Omicron) in adults ≥18 years of age | 14 days after a single dose of the booster vaccine
Cross-protecting effect of neutralizing antibodies against different variants (Alpha, Beta, Delta, and Omicron) in adults ≥18 years of age | 28 days after a single dose of the booster vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Khalifa Medical City, SEHA, Abu Dhab, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No